CLINICAL TRIAL: NCT01272856
Title: An Open-Label, Single-Center, Phase I Study on the Safety of Abatacept in Relapsing Polychondritis
Brief Title: Study on the Safety of Abatacept in Relapsing Polychondritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Stanford Peng, MD, Benaroya Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB10063
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Relapsing Polychondritis
MeSH Terms: conditions — Polychondritis, Relapsing | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Abatacept (Experimental)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — 125 mg pre-filled syringe for sub-q injection weekly.
  Other Names: Orencia

SUMMARY:
The purpose of this study is to test the safety of the study drug abatacept and see what effects (good and bad) it has in patients with relapsing polychondritis.

DETAILED DESCRIPTION:
After a screening period of up to 4 weeks, patients who fulfill all inclusion and exclusion criteria will receive open-label subcutaneous abatacept consisting of 125 mg weekly, beginning 1 week thru Week 24.

Throughout the study, blood will be collected for clinical laboratory safety, pharmacodynamics and biomarkers. Disease activity assessments will include laboratory evaluation of acute phase reactants, pulmonary function testing, computed tomography of the neck and chest, electrocardiogram, echocardiogram, audiogram, physician assessment of chondritis activity, swollen and tender joint counts, and patient- and physican-reported outcomes. Adverse events and concomitant medications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. Diagnosed with relapsing consisting of 2 major or 1 major + 2 minor criteria as follows:

   * Major criteria

     1. Proven inflammatory episodes involving auricular cartilage
     2. Proven inflammatory episodes involving nasal cartilage
     3. Proven inflammatory episodes involving laryngotracheal cartilage
   * Minor criteria

     1. Ocular inflammation (conjunctivitis, keratitis, episcleritis, uveitis)
     2. Hearing loss
     3. Vestibular dysfunction
     4. Seronegative inflammatory arthritis
   * Active RPC based on at least one of the following:

     * Active chondritis as defined as active inflammation, as observed by the Investigator, in auricular and/or nasal cartilage
     * Active tracheal and/or pulmonary disease documented by abnormal spirometry or chest computed tomography
   * Erythrocyte sedimentation rate ≥ 30 mm/hr or C-reactive protein ≥ 0.6 mg/dL
   * If receiving any of the following medications, has been on a stable dose for the durations indicated without intent to change throughout the study:

     * Azathioprine, methotrexate, mycophenolate, leflunomide: 1 month
     * Corticosteroids: 2 weeks
     * Nonsteroidal anti-inflammatory drugs (NSAIDs): 1 week
3. Age and Sex

   * Men and women, greater than 18 years of age
   * Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 10 weeks after the last dose of study drug to minimize the risk of pregnancy.

Women of child bearing age include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:

* Amenorrhea that has lasted for greater than 12 consecutive months without another cause, or
* For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.

Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or who are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.

Women of child bearing age must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of the investigational product.

A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study and for up to 10 weeks after the last dose of study drug to minimize the risk of pregnancy.

Exclusion Criteria:

1. Sex and Reproductive Status

   * Women of child bearing age who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 10 weeks after the last dose of study drug.
   * Women who are pregnant or breastfeeding.
   * Women with a positive pregnancy test on enrollment or before administration of abatacept.
2. Target Disease Exceptions

   * Fulfills American College of Rheumatology criteria for any other connective tissue disease, such as but not necessarily limited to systemic lupus erythematosus, systemic sclerosis (scleroderma), polymyositis or dermatomyositis, or rheumatoid arthritis, or possesses another distinct condition known to be associated with chondritis, such as Wegener's granulomatosis or Behcet's disease
   * Use of cyclophosphamide, cyclosporine A or tacrolimus within one month or at any time during administration of study drug
   * Use of biologic treatments within the timeframes indicated:

     * Anti-CD20 monoclonal antibodies or other immune cell-depleting therapy in the last 6 months or without evidence of appropriate lineage reconstitution
     * TNF antagonists, IL-1R antagonists, or co-stimulation modulators in the last 3 months
     * Any prior treatment with stem cell transplantation or other myeloablative therapy
   * Concomitant illness or disease activity which, in the opinion of the investigator, is likely to require significant additional immunosuppressive therapy (e.g. > 40 mg daily oral prednisone for asthma) during the course of the study
3. Medical History and Concurrent Diseases

   * Subjects who are impaired, incapacitated, or incapable of completing study-related assessments.
   * Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, whether or not related to RPC and which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
   * Female subjects who have had a breast cancer screening that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded by additional clinical, laboratory, or other diagnostic evaluations.
   * Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ. Existing non-melanoma skin cell cancers should be removed, the lesion site healed, and residual cancer ruled out before administration of the study drug.
   * Subjects who currently abuse drugs or alcohol.
   * Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of human immunodeficiency virus (HIV) detected during screening.
   * Subjects with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed.
   * Subjects who have received any live vaccines within 3 months of the anticipated first dose of study medication.
   * Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis, or bronchiectasis).
   * Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be subjects with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).
4. Physical and Laboratory Test Findings

   * Subjects must not be positive for hepatitis B surface antigen.
   * Subjects who are positive for hepatitis C antibody if the presence of hepatitis C virus was also shown with polymerase chain reaction or recombinant immunoblot assay.
   * Subjects with any of the following laboratory values

     * Hemoglobin < 8.5 g/dL
     * WBC < 3000/mm3 (< 3 x 109/L)
     * Platelets < 100,000/mm3 (< 3 x 109/L)
     * Serum creatinine > 2 times the ULN
     * Serum ALT or AST > 2 times the ULN
   * Any other laboratory test results that, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
5. Allergies and Adverse Drug Reactions

   * Known sensitivity to abatacept
6. Prohibited Treatments and/or Therapies

   * Subjects who have at any time received treatment with any investigational drug within 28 days (or less than 5 terminal half-lives of elimination) of the Day 1 dose.
   * Any concomitant biologic DMARD, such as anakinra.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 24 Weeks

SECONDARY OUTCOMES:
Physician assessment of chondritis burden | 24 Weeks
Acute phase reactants (ESR, CRP) | 24 weeks
Patient and physician-reported outcome measures, including HAQ, SF-36, and Visual Analogue Scores | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Peng SL, Rodriguez D. Abatacept in relapsing polychondritis. Ann Rheum Dis. 2013 Aug;72(8):1427-9. doi: 10.1136/annrheumdis-2013-203319. Epub 2013 Apr 20. No abstract available. PMID 23606702